CLINICAL TRIAL: NCT04080999
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation (r-TMS) Combined With Conventional Cognitive Treatment on Cognitive-behavioral Symptoms of Left Hemispatial Neglect in Right-stroke Patients Within Three Months Post-onset Compared to Conventional Cognitive Treatment Only: a Randomized Controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation in Spatial Attention After Stroke
Acronym: r-TMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Emanuela Casanova (Unknown); Francesco Di Gregorio (Unknown); Fabio La Porta (Unknown); Roberto Piperno (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17075
Record Dates: First submitted 2019-03-05; First posted 2019-09-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Stroke
Keywords: r-TMS; Hemispatial Neglect; Visual Scanning
MeSH Terms: conditions — Stroke; Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- r-TMS Group (Experimental): r-TMS Parameters International 10/20 system for the location of the target area (non-lesioned left parietal cortex) 60% Power Frequency: 1 Hz 90 pulse trains with 10 pulses each (total 900 stimuli), resulted in a total stimulation period of 15 minutes.
  Visual Scanning Visual-spatial training; Reading and copying training; Copying of line drawings on a dot matrix. Barrage
  Interventions: Device: r-TMS
- Sham Group (Sham Comparator): Sham stimulation and Visual scanning training
  Interventions: Device: SHAM

INTERVENTIONS:
Device: r-TMS — The interventions have a total administration time of 75 minutes per day.For TMS stimulation, the coil will be positioned tangentially on the target area. Each r-TMS session will last 15 minutes and will be administered every other day (e.g. Monday-Wednesday-Friday, Monday-Wednesday-Friday, Monday). The visual scanning treatment involves the presence of a therapist, who administers various visual scanning tasks, used to increase patient's awareness and to teach strategies to improve spatial exploration abilities (Pizzamiglio et al.,1992).Trainings include three increasing levels of difficulty (9 possible combinations). Each level of difficulty will be exercised until the patient reaches a level of accuracy of 75%. The CCT will be carried out in 50 minutes sessions for 5 days a week within 15 days (11 sessions in total). On the days when the r-TMS is also administered, the administration of the CCT will immediately follow the brain stimulation.
  Arms: r-TMS Group
Device: SHAM — Device: SHAM Stimulation and Visual Scanning training. In the control group, the coil of the r-TMS will be positioned at 90° on the target area, thus no specific cortical modulation will be implemented (SHAM stimulation). For the SHAM group, the CCT protocol will be administered with the same modalities and time frame as detailed for the intervention group.
  Arms: Sham Group

SUMMARY:
Randomized Controlled Trial (RCT) aiming at assessing the efficacy of a novel rehabilitation protocol, based on repetitive transcranial magnetic stimulation (r- TMS) in combination with a conventional cognitive treatment (CCT). The protocol will be statistically compared to the same CTT administered without the r-TMS in a sample of right-stroke patients (age between 18 and 80 years) with left hemispatial Neglect.

DETAILED DESCRIPTION:
BACKGROUND: A frequent and disabling impairment in persons who suffered acquired brain injury after stroke is left hemispatial neglect (LHSN). LHSN is a spatial attentive syndrome characterized by a reduced ability to attend, perceive and consciously represent the left contralesional space, in the absence of a primary sensory deficit. Commonly, the LHSN is due to a lesion on the right inferior parietal cortex and/or on the right fronto-parietal areas. Furthermore in stroke, LHSN is often associated with a mixture of attention and motor deficits leading to complex cognitive and behavioral pictures, which may even interfere with the administration of standard cognitive treatments for LHSN. However, several studies already demonstrated the efficacy of rehabilitation treatments on patients with LHSN, in terms of reducing disability, using various rehabilitative techniques and assessment tests. The rehabilitation techniques can be distinguished, accordingly to the used tools in: cognitive treatments (i.e. visual scanning training) and non-invasive brain stimulation methods (i.e. r-TMS). Conventional cognitive treatments (CCT) for LHSN involve different types of exercises aimed at reducing attentive bias for the ipsilesional space and/or promoting awareness of contralesional space by a continuous training of the patient's spatial exploration abilities. Instead, the TMS is a non-invasive method to modulate excitability of the cerebral cortex. The frequency of TMS pulse determines the type of modulation on the cerebral cortex (i.e. inhibitory <1 Hz; excitatory> 5 Hz). The most used TMS paradigm for the rehabilitation of LHSN is the r-TMS (repetitive transcranial magnetic stimulation) and it is based on the model of the inter-hemispheric competition. According to the model, the cerebral areas responsible for spatial orientation are contralateral to the attended hemifield (i.e. the left cerebral areas are responsible for the spatial orientation towards the right hemifield) and exert a reciprocal inter-hemispheric inhibition. The left and right fronto-parietal cortices are part of a intra-hemispheric network, which together with a parietal inter-hemispheric pathway, control the spatial orientation. In particular, a lesion on the right parietal cortex causes disinhibiting of the left parietal cortex and therefore a pathological over-activation of the latter.

According to the model, this left over-activation inhibits the right contralateral neural activity, as an increase of the healthy hemisphere inhibition activity on the damaged hemisphere. For these reasons, in the LHSN, a pathological orientation or pathological attention bias is determined towards the right hemifield after right stroke. Often, the r-TMS treatments aimed at rebalancing the inter-hemispheric competition through a stimulation of the parietal-parietal pathway, in particular inhibiting the intact areas of the left parietal cortex. The results showed significant post-treatment improvements in several neuropsychological and behavioral tests. In particular, a recent study showed how low- frequency r-TMS on the intact contralesional parietal areas reduced the clinical symptoms of LHSN after 10 treatment sessions. Improvements were stable 15 days after the treatment.

Despite evidence of efficacy of single treatment on cognitive symptoms of LHSN, many authors agree that the use of different rehabilitative techniques on the same patient are useful for generalizing clinical improvement and have a greater potential in reducing long-term global disability. However, in the literature, only few study tested effects of combined interventions on LHSN. Here, we aim at assessing the efficacy of a novel rehabilitation protocol, based on r-TMS in combination with a CCT, based on visual scanning training AIMS

To compare the efficacy of a combined r-TMS and CCT intervention aiming at reducing cognitive symptoms of LHSN, in a sample of right Stroke patients with LHSN, within the context of an RCT.

To evaluate the long- term impact of the intervention To evaluate the effect of the intervention on other clinical measures (activity of daily living, attentive and motor functions) and on psychophysiological indices.

METHODS: Multicenter, Randomized Controller Trial, with blind assessments on pre-test, post-test and on 3 months follow-up.

POPULATION: Right stroke patients with clinical evidence of LHSN INTERVENTION: Inhibitory low-frequency r-TMS on the intact left parietal cortex combined with a conventional cognitive treatment (visual scanning training) for 2 weeks. Multidisciplinary assessment with clinical and psychophysiological indices.

CONTROL: SHAM group with a placebo r-TMS stimulation combined with visual scanning training for 2 weeks. Multidisciplinary assessment with clinical and psychophysiological indices.

OUTCOMES:

The primary outcome is represented by a specific assessment of cognitive symptoms in LHSN with the Behavioral Inattention Test (BIT)

The secondary outcomes will consider the impact of the intervention on other clinical and psychophysiological indices. In particular we will test:

Activity of daily living and everyday life independence, attentive functions and motor independence.

A psychophysiological index based on Visual-Evoked Potentials

(VEPs). In particular we will focus on the N1 component, a posterior negativity, which is altered in terms of latency and amplitude in LHSN population. In order to study effects of the r-TMS in the inter-hemispheric parietal pathway, we will extract indices of inter-hemispheric transmission time (IHTT) on the N1 latency and of spatial attention bias on N1 amplitude.

EXPECTED RESULTS: In the intervention and in the control groups we expect a significant improvement of the clinical (cognitive, activity of daily living, attentive and motor functions) and psychophysiological indices, because both groups will be treated with an effective rehabilitation protocol (visual scanning training).

However, unlike the standard methods of rehabilitation, the new techniques of magnetic stimulation such as r-TMS allow the execution of a cognitive task through the pre-empowerment of a specific network or neuronal circuit. This effect could facilitate experiential learning during cognitive training, with a richer and more articulated neural environment, as well as selectively stimulated according to the areas most involved in the lesion. In the case of LHSN the mechanism of empowerment concerns the preserved parietal areas and the inter-hemispheric connectivity. As a consequence, r-TMS could increase the "responsiveness" of the peri-lesional areas and of the inter- hemispheric connectivity during cognitive training, increasing its effectiveness with respect to the SHAM condition. Therefore, we expect a larger improvement on the intervention group, because the r-TMS could modulate the responsiveness of the specific spatial attention pathway. At three months, it is expected a stabilization of functional improvements.

Randomization method In order to ensure that each arm will contain an equal number of individuals, eligible subjects will be randomly assigned to one of the two groups with a blocked randomization method based on a block size of 4.

Assessor and patient blindness: obviously, the physician who will administer the r- TMS or the SHAM stimulation will not be blind to the randomization. However, to ensure a double-blind assessment, pre-treatment assessments will be performed prior to randomization. An assessor not aware of the patient randomization group will conduct post-treatment and follow-up assessments. Also the visual scanning protocol will be administered by therapists unaware of the patient randomization and patients themselves will be instructed not to reveal any information on the brain stimulation treatment received.

Case report form and data monitoring Specific case report forms (CRF) for every test in the assessments are already available and will be used. During the treatment the responsible physician will report any adverse event in the treatment-CRF. All information and results will be promptly reported on the electronic database. A researcher will be responsible for the electronic database, data analyses and will draft the single patient record at the end of all procedures.

Maximization of inter-rater reliability of assessment and treatment methods

In order to minimize biases deriving from inter-rater measurement errors, the following interventions will take place during the start-up stage:

1. Collegial assessment of voluntary patients by the various assessors and therapists in order to standardize the administration modalities and resolve discrepancies between scoring and treatment procedures.
2. Subsequent development of an "assessment manual" and of a "treatment manual" containing all information necessary to the administering and scoring procedures.

Cases lost at follow-up In case of lost to follow-up, the information available up to that moment will be considered. If participant is lost at follow-up, it will be analyzed on the basis of the "intention to treat" principle. Finally, the reason for quit the study will be reported for each participant lost at follow-up.

Sample size

The sample size was calculated using the following formula:

https://www.dropbox.com/s/y56umrt7z93en1w/Simple%20size%20formula.docx? dl=0

The sample size resulting from the formula calculated for the BIT is 25.2. Consequently, the minimum sufficient simple to reach the primary aim is, assuming approximately 10% of subjects lost to follow-up, 60 subjects (30 X group) recruited over a three-year period.

Data Analyses In order to evaluate cognitive symptoms of LHSN in the two groups (primary outcome), differences in the BIT will be analyzed, between the pre-treatment (T0), post-treatment (T1) and follow-up (T2) phases for both groups of patients (r-TMS + CCT group and SHAM + CCT group). For this purpose, analyses of covariance will be performed for the BIT scale using a mixed-model ANCOVA with a 2X3 design, where the "between" factor is represented by the randomization group (r-TMS + CCT, SHAM + CCT) and the "within" factor is represented by the assessment time (T0, T1, T2). Whenever necessary, Greenhouse-Geiser correction will be applied and corrected p-values will be reported. In the ANCOVA, an adjustment will be made for the pre-treatment values and other possible confounding factors such as age, gender and education of the participants. Besides p-values, effect sizes will be provided in order to assess the size of treatment effect. Similar analyses will be performed also for the secondary outcomes on clinical and psychophysiological measures. Data analysis will be performed using Matlab (The Mathworks Inc.) and SPSS (version 13).

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of ischemic stroke in the right middle cerebral artery or right intra-cerebral hemorrhagic stroke, confirmed by brain CT and / or brain MRI;
2. Diagnosis of LHSN with a specific test (asymmetry score on Bells cancellation test > 3]);
3. Intra-hospital rehabilitation setting (ordinary hospitalization or DH) or outpatient setting;
4. Age between 18 and 80 years;
5. Time between stroke onset and study recruitment three weeks to three months;
6. Availability to provide informed consent to participation.

Exclusion criteria

1. Clinical instability at recruitment (for example, fever, acute internist conditions, etc.);
2. History of epilepsy and / or occurrence in the acute phase of at least one seizure crisis
3. Presence of intracranial metallic implants;
4. Presence of devices, which could be altered by r-TMS, such as pacemakers, ventricular-peritoneal derivations, Baclofen pump;
5. Absence of a bone operculum following a neurosurgical operation of decompressive craniotomy;
6. Presence of behavioral disturbances with inversion of the sleep-wake rhythm
7. Mono- or bilateral occipital lesions documented on CT and / or history of cortical blindness or visual agnosia;
8. Concomitant psychiatric disorders and / or history of substance abuse;
9. State of pregnancy
10. Inability to execute the following simple order: "Take the pen instead of the key and put it on the sheet"
11. Severe acoustic deficit not corrected by the use of a hearing aid
12. Severe reduction of the visus despite the use of eyeglasses
13. Positive anamnesis of previous cognitive decline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline: behavioral Inattention Test (BIT) | up to 21 days post baseline and up to 90 days follow-up
  A battery for the assessment of cognitive and behavioral symptoms in LHSN

SECONDARY OUTCOMES:
Change from Baseline: catherine Bergegò Scale (CBS) | up to 21 days post baseline and up to 90 days follow-up
  A battery for the assessment of LHSN symptoms in the activity of daily living.
Change from Baseline: test of Attention Performance (TAP/TEA) | up to 21 days post baseline and up to 90 days follow-up
  two subtest will be executed "alertness" and "Visual field/Neglect" to assess attentive functions
Change from Baseline: functional independence measure (FIM) | up to 21 days post baseline and up to 90 days follow-up
  The motor subscale will be executed to assess motor independence
Change from Baseline: Motricity Index (MI) | up to 21 days post baseline and up to 90 days follow-up
  A test to assess motor impairment in stroke patients.
Change from Baseline: Trunk Control Test (TCT) | up to 21 days post baseline and up to 90 days follow-up
  A test to assess the ability to control the trunk after stroke.
Change from Baseline: Inter Hemispheric transmission Time (IHTT) | up to 21 days post baseline and up to 90 days follow-up
  Psychophysiological index of inter-hemispheric transmission.
Change from Baseline: visual-Attention Bias Index (vABI) | up to 21 days post baseline and up to 90 days follow-up
  Psychophysiological index of inter-hemispheric imbalance in a visual-spatial attention task

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Maggiore, Bologna, Bo
  - Azienda Unità Sanitaria Locale, Bologna

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data for all primary and secondary outcome measures will be made avalaible
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963
- [Derived] Di Gregorio F, La Porta F, Casanova E, Magni E, Bonora R, Ercolino MG, Petrone V, Leo MR, Piperno R. Efficacy of repetitive transcranial magnetic stimulation combined with visual scanning treatment on cognitive and behavioral symptoms of left hemispatial neglect in right hemispheric stroke patients: study protocol for a randomized controlled trial. Trials. 2021 Jan 6;22(1):24. doi: 10.1186/s13063-020-04943-6. PMID 33407787
- See also: Azouvi, P., Jacquin-Courtois, S., & Luauté, J. (2016). Rehabilitation of unilateral neglect: Evidence-based medicine. Annals of Physical and Rehabilitation Medicine. — http://doi.org/10.1016/j.rehab.2016.10.006
- See also: Barnett, K. J., & Corballis, M. C. (2005). Speeded right-to-left information transfer: The result of speeded transmission in right-hemisphere axons? Neuroscience Letters, 380(1-2), 88-92. — http://doi.org/10.1016/j.neulet.2005.01.025
- See also: Corbetta M, Kincade MJ, Lewis C, Snyder AZ, & A., S. (2005). Neural basis and recovery of spatial attention deficits in spatial neglect. Nat Neurosci., 8(11), 1603-1610 — http://doi.org/10.1038/nn1574
- See also: Di Russo, F., Bozzacchi, C., Matano, A., & Spinelli, D. (2013). Hemispheric differences in VEPs to lateralised stimuli are a marker of recovery from neglect. Cortex, 49(4), 931-939 — http://doi.org/10.1016/j.cortex.2012.04.017
- See also: Dietz, M. Et:al., (2014). Effective connectivity reveals right-hemisphere dominance in audiospatial perception: implications for models of spatial neglect. The Journal of Neuroscience : The O — http://doi.org/10.1523/JNEUROSCI.3765-13.2014
- See also: Jacquin-courtois, S. (2015). ScienceDirect Hemi-spatial neglect rehabilitation using non-invasive brain stimulation : Or how to modulate the disconnection syndrome ? Annals of Physical and Rehabilitation Medicine, 58(4), 251-258. — http://doi.org/10.1016/j.rehab.2015.07.388
- See also: Müri, R. M., Cazzoli, D., Nef, T., Urs, P., & Nyffeler, T. (2013). Non-invasive brain stimulation in neglect rehabilitation : an update, 7(June), 1-10. — http://doi.org/10.3389/fnhum.2013.00248
- See also: Oliveri, M. (2011). Brain stimulation procedures for treatment of contralesional spatial neglect. Restorative Neurology and Neuroscience. — http://doi.org/10.3233/RNN-2011-0613
- See also: Sozzi, M., Balconi, M., Arangio, R., Pisani, L., & Mariani, C. (2012). Top-down strategy in rehabilitation of spatial neglect: How about age effect? Cognitive Processing, 13(1 SUPPL), 339-342 — http://doi.org/10.1007/s10339-012-0493-5